CLINICAL TRIAL: NCT03049904
Title: American Indian and Alaska Native Men Who Have Sex With Men HIV & Substance Abuse Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karina Walters, Associate Dean for Research; William P. and Ruth Gerberding Endowed University Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00000597; 5K24DA031613 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-10 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: HIV; Substance Use
Keywords: Indian, North America; Male, Two-Spirit; HIV Prevention; MSM
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List Control (No Intervention): Participants wait 3 weeks before receiving the intervention.
- Experimental Vr2L 2Spirit (Experimental): Participants immediately begin their participation in the virtual world.
  Interventions: Behavioral: Vr2L 2Spirit

INTERVENTIONS:
Behavioral: Vr2L 2Spirit — Three weeks exploring the Vr2L 2Spirit island.
  Week 1: Learning Level. Contains the Vr2L 2Spirit island orientation, the learning paths covering HIV testing, harm reduction, safer sex, and condom use & condom use negotiation, the lodge, the in-world Motivational Interviewing (MI) counseling, and leisure activities.
  Week 2: Skills Building Level. The purpose of the city level is for participants to practice the knowledge gained in the Learning level through quests, challenges, and role play scenarios.
  Week 3: Experiential Level. Experiential interactions with other participants where they can practice the knowledge and skills they gained in the previous levels.
  Arms: Experimental Vr2L 2Spirit

SUMMARY:
This is a pilot study of the feasibility of the virtually reality, online, culturally grounded HIV prevention intervention for Native American men who have sex with men. The project will include 90 Native American men who have sex with men (MSM) from across the continental United States as well as Alaska and Hawaii.

The investigators will use a randomized clinical trial with a waitlist control condition to evaluate the intervention's impact on HIV / Sexually Transmitted Infections (STI) testing behavior, condom use, and substance use harm reduction. Specifically, investigators will ask participants to spend 3 weeks exploring a virtual reality environment hosted in the Second Life® platform. The island consists of 3 levels: Learning Level, Skills building level, and Experiential level.

In the Learning level the participant's avatar will have the opportunity to attend up to 2 free Motivational Interviewing sessions to establish their goals for their time on the island. Additionally, they will explore 4 learning paths each covering a knowledge objective: HIV Testing, Condom Use & Condom Use Negotiation, Safer Sex, and Harm Reduction. Each path will present knowledge via videos, interactive games, stories, and teachings. After completing level 1, participants will move on to the Skills building level. Here participants will have the opportunity to role play scenarios (e.g., obtaining an HIV test, requesting PrEP from their doctor, negotiating condom use) with pre-program virtual actors. All scenarios are based on the knowledge gained in the Learning Level. Participants will also engage on mini-quests for additional knowledge and in-world rewards. Finally, in the third level participants will be able to practice the skills learned in interactions with other participants' avatars.

If efficacious, this online HIV prevention intervention has the potential for widespread dissemination and could be particularly helpful for rural and reservation-based Native MSM who often have difficulty accessing services and support.

DETAILED DESCRIPTION:
Recruitment

Recruitment is nationwide via online ads in Gay, Bisexual, Trans, and Questioning (GBTQ) dating sites such as Grindr, GROWLr, Jack'd, etc. Investigators will send emails and flyers to partners in GBTQ and Two-Spirit organizations for them to advertise within their listservs and centers. Finally, investigators and project consultants will reach out to other researchers and community partners asking them to advertise the project within their own communities and organizations. Investigators expect a certain amount of "word-of-mouth" recruitment to occur as well.

Screening

* Participants are screened over the phone using a screening script.
* Men who screen out will be given a community resource list either by mail or email.
* If a person is eligible, but declines to participate, they will be given a brief one item exit question regarding general reason for nonparticipation.
* If needed, participants are walked through the process of creating a free Second Life® (SL) account and downloading the SL software onto their computer.

Online Consent

An email is sent to the participant with consent information and baseline assessment links. Prior to beginning the baseline assessment in REDCap, participants will read and confirm their consent (click "I agree to participate" or "I do not wish to participate"). Once participants consent online, they are assigned a study survey ID number and take the baseline assessment.

Assessments

The assessment is conducted via Research Electronic Data Capture (REDCap) a mature, secure web application for building and managing online surveys and databases. After completing the baseline assessment, participants are randomly assigned to either the Immediate or the 3-week Waitlist group. Participants in the immediate group will be asked to complete 3 online assessments (Baseline, end of intervention, and 3-month follow up). Participants in the Waitlist group will be asked to complete 4 an additional assessment at the end of their wait period. Participants will be paid in Tango gift cards for each survey completed.

IMMEDIATE participants. After completing the Baseline assessment, they will receive an email containing: their Tango card information, the invitation to the private island, their unique Personal Identification Number (PIN) for accessing the private island as well as a Second Life® How-to guide and a community resource list.

WAITLIST participants. After completing the baseline assessment, they will enter a 3-week wait period. At the end of the 3-week wait period, they complete the Baseline 2 (End of waitlist) survey in REDCap. They will then proceed through the same steps as the Immediate group.

Intervention

The intervention in the Virtual Two Spirit (Vr2L 2Spirit) project is conducted exclusively online through the SL® platform. SL is a free and 3-dimensional online virtual world developed by Linden Lab.

Accessing the Vr2L 2Spirit Island

SL® consists of both public and private virtual spaces. The Vr2L 2Spirit island is a private island and only those avatars who have been authorized access by study staff are able to find it and enter it. Participants cannot grant access to other people.

The Vr2L 2Spirit island.

The island is split into three levels: 1) learning paths, 2) skill building, and 3) experimental. Access to the levels are locked hierarchically, meaning that until participants complete a lower level they will not gain access to the higher levels; however, once they successfully complete a level they are welcomed to return to it as often as they like. Participants are expected to complete each level in approximately one week; although they are allowed to complete it sooner and some may take a bit longer. We will encourage participants to move through the intervention in 3 weeks. Participants will be paid in Tango gift cards for each level completed whether they complete it in 2 days or in two weeks. If necessary, staff will use reminder emails, texts, in-world messages, and phone calls to encourage participants to complete the level in the allotted time.

Participants will be informed that their avatars' actions, interactions, and conversations with the programmed scenarios and with other avatars are considered data, and will be analyzed as part of the research study.

Level 1 - The Learning Level: 1st Week.

1. Orientation. After the participants' avatar authentication is completed, they will teleport to the orientation caves. Here they will receive a brief orientation to the Vr2L 2Spirit island and a refresher on basic SL skills needed to successfully navigate the virtual experience. Afterward they are free to explore the Vr2L 2Spirit island.
2. In-World Counseling. Participants will have the option of receiving up to two free Motivational Interviewing (MI) counseling sessions in the Vr2L 2Spirit island with an MI trained counselor. The counseling sessions will be confidential and will be an opportunity for participants to discuss their goals during their participation in this study.
3. Learning Paths. The main component of level 1 is the learning paths. There are 4 learning paths that cover different areas of HIV prevention: safer sex, harm reduction, condom use, and HIV testing. Each learning paths consists of some combination of videos, scripted interactions, interactive exercises, and small quests or games.

   1. Safer sex. Includes information on Pre-Exposure Prophylaxis (PrEP): what it is, how to use it, and how to obtain it. It also covers the risks of sexual intercourse with multiple partners and ways participants can protect themselves and their partners. Additionally, it covers strategic positioning, sero-sorting and its risks. Finally, it addresses partner's behavior and ways in which the participant can protect themselves and their partner.
   2. Harm reduction. Includes a definition of harm reduction, information on how one can reduce harm from IDU, other substances, and binge drinking. Finally, it addresses how to decrease IDU risk of HIV exposure.
   3. Condom use / condom negotiation. Includes information on the different types of condoms, how to use them, and how to bring up and negotiate condom use with your partner.
   4. HIV Testing. Includes information on types of HIV tests, where to find testing sites, the testing experience, and what happens after your HIV results are back.

   While walking the paths, learning participants will have the opportunity to collect traditional medicines or materials (e.g., corn, prairie sage, birch bark, flowering tobacco). These collectibles can be turned into the lodge where the participant will learn about the traditional uses of these materials.

   As participants move through the learning paths, they will gain in-world coins for completing tasks. The coins gained in the Vr2L 2Spirit island are specific to the Vr2L 2Spirit island only. Participants can use these coins to purchase in-world rewards such as additional customization for their avatar (e.g., clothing, hats, accessories, tattoos).
4. The Lodge. It contains the MI counseling rooms, a smudging station, the collectibles station, the store containing avatar accessories (e.g., clothing, hats, sunglasses, jewelry). There is also a receptionist available to answer participants' questions.
5. Leisure activities. Level 1 also contains many opportunities for leisure activities such as horseback riding, canoeing, wind surfing, drum circle and a camp fire among others. These activities are not a required portion of the interaction and are instead created to enhance the immersion experience, provide fun and relaxation alongside the learning experience, and allow for participants to build camaraderie with their fellow participants.

Level 2 - The City Level: 2nd Week.

The city level or skill-building level contains the clinic, the park, the bookstore, the Q-center, the nightclub, and the city store. The purpose of the city level is for participants to practice the knowledge gained in level 1 through quests, challenges, and role-play scenarios.

1. Challenges. There are six city challenges created to reinforce participants' knowledge. All challenges must be completed before gaining access to the Level 3 - Bathhouse.

   1. HIV Test. In the clinic, the avatar will have the opportunity to take a Rapid Response HIV test at the clinic. The participant will have the option of selecting their avatar's HIV status or be randomly assigned an HIV status after taking the test.
   2. PrEP. If HIV negative, avatar will have the option of requesting a prescription for Pre-Exposure Prophylaxis (PrEP) at the city clinic. Participants will receive counseling regarding PrEP and will be able to purchase the PrEP prescription at the city store.
   3. Condoms. Avatars will be required to pick up free latex condoms at the city clinic. They also have the option of purchasing polyurethane, polyisoprene, or sheepskin condoms at the city store.
   4. Needle exchange. Avatars will be required to find a dirty needle in the city and exchange it for a clean needle at the clinic. Using the dirty or clean needle is not required.
   5. Book challenge. Hidden around the city landscape are six books. Every time an avatar finds a book, they are given a fact related to HIV prevention.
   6. Role play scenarios. More information below.
2. Role play scenarios. Throughout the city participants will encounter a series of role-play scenarios related to harm reduction, safer sex, condom use, and HIV testing. The role-plays are scripted; however, they allow participants to make decisions throughout the interactions which will allow them to experience likely outcomes based on their choices. In order to move on to level 3, they must complete each scenario at least once.

   1. Drug use. This role-play will allow participants to practice the skills around harm reduction with intravenous drug use (IDU).
   2. Anonymous / Casual sex. This role-play allows the participant the opportunity to practice skills around anonymous / casual sexual intercourse.
   3. Binge drinking. This role-play allows the participant the opportunity to practice skills around harm reduction related to binge drinking.
   4. Condom use. This role-play allows the participant the opportunity to practice skills around condom use and condom use negotiation.
   5. Teaching opportunity. This role-play allows the participant the opportunity to assume the role of teacher. They will encounter a younger Native American man who has questions about the four content areas. The participant will have the opportunity to answer the stranger's questions thus reinforcing their own knowledge.
   6. HIV Testing. This role-play scenario allows the participant to gain further knowledge about the HIV testing experience.
3. At the end of level 2. After completing all the city challenges, participants are granted access to Level 3 - Experiential.

Level 3 - The Experiential Level: 3rd Week.

Physically located in the city space of the Vr2L 2Spirit island, the area is nevertheless locked to participants until they complete all the challenges on level 2. Once participants have gained access, they will be in a "free play" area; although their interactions are still monitored and recorded. The participants is reminded of this through signage upon entering the locker room. There are no scripted interactions in this space. Interactions will be limited to other participants' avatars only.

End of Intervention Assessment Debrief Phone Call

On the next business day after the participant has completed one-week in Level 3 , they will receive the prompt to take the next online survey in REDCap.

Participants will also be contacted to schedule a debriefing interview with study staff. Participants will be asked debriefing questions about their experience in the virtual world.

Three Month Follow-up Assessment

Approximately three months after the participant completes Level 3 of the island, they will receive an email asking them to complete the final (follow-up) survey.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Self-identified as American Indian or Alaska Native
* Either: enrolled in their Tribe; eligible for enrollment in their Tribe; OR at least ¼ blood quantum (across all tribes).
* Male (assigned "male" gender at birth or assigned "female" gender at birth but now identify as "male")
* Have access to a computer with internet access and the ability to download the Second Life® software.
* Reside within the United States of America
* Have engaged in sexual intercourse with a man in the previous 3 months.
* Have used substance (drugs or alcohol) in the previous 3 months.
* Either unknown HIV status or HIV negative.

Exclusion Criteria:

* Suicidal ideation, plan, or attempt in the previous 2 weeks.
* Women
* Younger than 18 years old
* Non-Native American

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned "male" gender at birth or assigned "female" gender at birth but now identify as "male"
Enrollment: 79 (Actual)
Dates: Start 2017-02-19 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Drug Use as assessed by Phen-X Toolkit for 30-Day Use | Baseline and Post Intervention (1 month); Baseline and 3 month Follow-up
  This measure can be used to assess the participant's recent consumption of a substance.
Change in Alcohol Use as assessed by Alcohol Use Disorders Identification Test (AUDIT) | Baseline and Post Intervention (1 month); Baseline and 3 month Follow-up
  Screening test developed for measuring excessive drinking.
Change in High Risk Sexual Behavior as assessed by National Institute on Drug Abuse (NIDA) HIV Risk Behavior questionnaire | Baseline and Post Intervention (1 month); Baseline and 3 month Follow-up
  Survey that measures injection and sexual risk behaviors for contracting HIV.
Change in HIV Testing behavior as assessed by STI / HIV Testing Self Efficacy | Baseline and Post Intervention (1 month); Baseline and 3 month Follow-up
  Survey that measures changes in confidence regarding STI and / or HIV testing behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Karina L Walters, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No